CLINICAL TRIAL: NCT05682885
Title: The Effectiveness of Lymphatic Bypass Supermicrosurgery for Primary Lymphedema Prevention After Breast Cancer Axillary Lymph Node Dissection: a Randomized Controlled Study
Brief Title: The Effectiveness of Lymphatic Bypass Supermicrosurgery
Acronym: ELYBS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dharmais National Cancer Center Hospital (Other Government)
Responsible Party: Principal Investigator, Bayu Brahma, Principal Investigator, Dharmais National Cancer Center Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 227/KEPK/IX/2022
Record Dates: First submitted 2022-11-22; First posted 2023-01-12 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Related Lymphedema; Lymphedema Arm
Keywords: Lymphatic Bypass Supermicrosurgery; Primary Lymphedema Prevention; Axillary Lymph Node Dissection
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: This study is a single-blind pragmatic parallel arm randomized clinical trial to analyze the effectiveness of lymphatic bypass supermicrosurgery (LBS).
Who Masked: Participant
Masking Description: Blinding is implemented in two conditions: the main researcher (Bayu Brahma) will not know the identity and medical history of the patient when assessing the indocyanine green (ICG) lymphography results and the patients will not know the received type of surgical procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Axillary lymph node dissection with LBS (Experimental): 70 subjects will be needed for each group. A standard mastectomy or lumpectomy incision is made and ALND will be done in the same incision. The lymphatic vessels and lymph nodes will be resected using a near-infrared (NIR) camera. To locate lymphatic vessels, a microscope with ICG lymphography navigation is employed. LBS was performed by making intima-to-intima anastomosis between the afferent lymphatic vessels and the recipient's veins, or to the efferent lymphatic vessels. The anastomosis patency will be assessed by observing the ICG fluorescent flow. After surgery, follow-up will be done every 2 months and every 3 months in the second year. UEL index, ICG lymphography, and quality of life evaluation will be done. The cumulative incidence of BCRL, the free survival time of BCRL, and subclinical lymphedema (SCL) progression will be reported descriptively. BCRL risk factors and collateral lymphatic pathway will be observed as well.
  Interventions: Procedure: Lymphatic Bypass Supermicrosurgery
- Axillary lymph node dissection without LBS (No Intervention): 70 subjects will be needed for each group. A standard mastectomy or lumpectomy incision is made and ALND will be done in the same incision. After primary breast cancer removal, a standard ALND level I, II, and if necessary, level III is performed. After surgery, follow-up will be done every 2 months and every 3 months in the second year. History taking, physical examination, radiology and histopathology examination, UEL index, and ICG lymphography evaluation will be done during follow-up. Each subject will complete the lymphedema quality of life questionnaire. The cumulative incidence of BCRL, the free survival time of BCRL, and SCL progression will be reported descriptively. BCRL risk factors and collateral lymphatic pathway will be observed as well.

INTERVENTIONS:
Procedure: Lymphatic Bypass Supermicrosurgery — Axillary Lymph Node Dissection with Lymphatic Bypass Supermicrosurgery
  Arms: Axillary lymph node dissection with LBS

SUMMARY:
This study evaluate the effectiveness of lymphatic bypass supermicrosurgery (LBS) and axillary lymph node dissection (ALND) compare to ALND alone to prevent breast cancer treatment-related lymphedema (BCRL).

DETAILED DESCRIPTION:
In the intervention group, LBS was performed after ALND with the intima-to-intima coaptation using the supermicrosurgery technique. The anastomosis is done between the afferent lymphatic vessel to the recipient's vein, or if possible, from the afferent to the efferent lymphatic vessel. The upper extremity lymphedema (UEL) index and indocyanine green (ICG) lymphography are utilized to evaluate the development of lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patient aged >18 years old
* Breast cancer patient with clinically ALNs metastases (cN1 or cN2).
* Breast cancer patient with no clinical metastasis and tumor size ≥5cm or no sentinel lymph node biopsy facility in the hospital.
* Any breast cancer patients that receive neoadjuvant systemic therapy.

Exclusion Criteria:

* Stage IV breast cancer patients who do not show clinical and radiological improvement after primary systemic therapy.
* Breast cancer patients with previous surgeries such as mastectomy, axillary lymph node biopsy, sentinel lymph node biopsy (SLNB), and ALND.
* Breast cancer patients with prior breast, chest wall, axillary, or neck radiotherapy.
* Breast cancer patients with preoperative lymphatic system abnormality detected by ICG lymphography.
* Breast cancer patients with iodine allergy, asthma, decreased kidney function, pregnancy, and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-11-18 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of BCRL | 1 year
  BCRL definition:
  Post operation subject condition with presence of minimum DB 2 with one or both symptoms (swelling, heaviness), and increment of UEL index >10% compared to pre operation
  OR
  Post operation subject condition with presence of ≥ DB 2 with minimum area 30% in one arm region in one of the arm lymphatic pathway (anterior or posterior), without presence of symptoms (swelling or heaviness), and increment of UEL index >10% compared to pre operation

SECONDARY OUTCOMES:
BCRL and SCL progression-free survival rate | 1 year
  Percentage of subjects who do not progress to subclinical lymphedema or lymphedema during the research.
Collateral lymphatic pathway | 1 year
  The number of lymphatic pathways flow into the region: supraclavicular, internal mammary, and contralateral axillary and supraclavicular nodes based on the ICG lymphography.
Quality of life lymphedema | 1 year
  Assessment of lymphedema quality of life score after the surgery using the lymphedema quality of life score questionnaire that is self-reported by the subjects every 2 months and every 3 months in the second year. Calculation of the lymphedema quality of life score is the summation of the score from each question. The minimum score is 0 and the maximum score is 100. A higher score indicates lower lymphedema quality of life.

OTHER OUTCOMES:
Association of body mass index (BMI) with BCRL | 1 year
  BMI was calculated by weight (kilograms) and height (centimeters). Categorized based on Asia Pacific classification are overweight (BMI ≥ 23 kg/m^2) and no overweight (BMI < 23 kg/m^2). Measured at one time point.
Association of number of axillary lymph nodes metastases with BCRL | 1 year
  The number of metastases lymph nodes and classified into >3 lymph nodes and ≤3 lymph nodes. Measured at one time point.
Association of number of taxane chemotherapy with BCRL | 1 year
  Taxane chemotherapy data from the subject's medical record and categorized into yes or no. Measured at one time point.
Association of regional lymph node radiation with BCRL | 1 year
  Regional lymph node radiation data from the subject's medical record and categorized into yes or no. Measured at one time point
Association of axillary fat weight with BCRL | 1 year
  Axillary fat weight in grams is taken at the time of surgery. Measured at one time point.

CONTACTS AND LOCATIONS:
Overall Officials: Bayu Brahma, MD, Principal Investigator — Dharmais Hospital National Cancer Center, Indonesia
Locations (1):
- Dharmais National Cancer Center Hospital, Jakarta, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be shared. The researcher provides a methodologically sound proposal. The proposal should be directed to bbrahma@dharmais.co.id. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 3 years following article publication.
Access Criteria: Qualified researchers who have received principal investigator's approval.

REFERENCES:
- [Background] Brahma B, Yamamoto T. Breast cancer treatment-related lymphedema (BCRL): An overview of the literature and updates in microsurgery reconstructions. Eur J Surg Oncol. 2019 Jul;45(7):1138-1145. doi: 10.1016/j.ejso.2019.01.004. Epub 2019 Jan 4. PMID 30638810
- [Background] Brahma B, Putri RI, Reuwpassa JO, Tuti Y, Alifian MF, Sofyan RF, Iskandar I, Yamamoto T. Lymphaticovenular Anastomosis in Breast Cancer Treatment-Related Lymphedema: A Short-Term Clinicopathological Analysis from Indonesia. J Reconstr Microsurg. 2021 Oct;37(8):643-654. doi: 10.1055/s-0041-1723940. Epub 2021 Mar 1. PMID 33648010
- [Background] Yamamoto T, Yamamoto N, Doi K, Oshima A, Yoshimatsu H, Todokoro T, Ogata F, Mihara M, Narushima M, Iida T, Koshima I. Indocyanine green-enhanced lymphography for upper extremity lymphedema: a novel severity staging system using dermal backflow patterns. Plast Reconstr Surg. 2011 Oct;128(4):941-947. doi: 10.1097/PRS.0b013e3182268cd9. PMID 21681123
- [Background] Yamamoto T, Narushima M, Yoshimatsu H, Yamamoto N, Kikuchi K, Todokoro T, Iida T, Koshima I. Dynamic Indocyanine Green (ICG) lymphography for breast cancer-related arm lymphedema. Ann Plast Surg. 2014 Dec;73(6):706-9. doi: 10.1097/SAP.0b013e318285875f. PMID 24322632
- [Background] Brahma B, Putri RI, Karsono R, Andinata B, Gautama W, Sari L, Haryono SJ. The predictive value of methylene blue dye as a single technique in breast cancer sentinel node biopsy: a study from Dharmais Cancer Hospital. World J Surg Oncol. 2017 Feb 7;15(1):41. doi: 10.1186/s12957-017-1113-8. PMID 28173818
- [Background] Akita S, Nakamura R, Yamamoto N, Tokumoto H, Ishigaki T, Yamaji Y, Sasahara Y, Kubota Y, Mitsukawa N, Satoh K. Early Detection of Lymphatic Disorder and Treatment for Lymphedema following Breast Cancer. Plast Reconstr Surg. 2016 Aug;138(2):192e-202e. doi: 10.1097/PRS.0000000000002337. PMID 27465179
- [Background] Ishiura R, Yamamoto T, Saito T, Mito D, Iida T. Comparison of Lymphovenous Shunt Methods in a Rat Model: Supermicrosurgical Lymphaticovenular Anastomosis versus Microsurgical Lymphaticovenous Implantation. Plast Reconstr Surg. 2017 Jun;139(6):1407-1413. doi: 10.1097/PRS.0000000000003354. PMID 28538568
- [Background] Yamamoto T, Yamamoto N, Hara H, Mihara M, Narushima M, Koshima I. Upper extremity lymphedema index: a simple method for severity evaluation of upper extremity lymphedema. Ann Plast Surg. 2013 Jan;70(1):47-9. doi: 10.1097/SAP.0b013e3182275d23. PMID 21734534
- [Background] Suami H. Anatomical Theories of the Pathophysiology of Cancer-Related Lymphoedema. Cancers (Basel). 2020 May 23;12(5):1338. doi: 10.3390/cancers12051338. PMID 32456209